CLINICAL TRIAL: NCT02708147
Title: Impact of Respiratory Physiotherapy in Children With Bronchiolitis in the First Two Years of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aveiro University (Other)
Responsible Party: Principal Investigator, Alda Sofia Pires de Dias Marques, Senior Lecturer, Aveiro University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PhDPT/VeronicaAbreu/2016
Record Dates: First submitted 2016-03-09; First posted 2016-03-15 (Estimated); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Bronchiolitis
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional treatment (Sham Comparator): Conventional treatment means that there will be only contact with physician/paediatrician and maybe drugs prescription.
  Only evaluations will be made at baseline and on the 3th, 5th and 21st days and an interview 30 days after.
  Interventions: Other: Conventional treatment
- Physiotheraphy + Conventional treatment (Experimental): Apart Conventional treatment a Physiotherapy protocol (techniques and education) will be performed on 5 sessions and evaluations will be made after each session as well as on baseline and on the 3th, 5th and 21st days and an interview 30 days after.
  Interventions: Other: Physiotheraphy + Conventional treatment

INTERVENTIONS:
Other: Physiotheraphy + Conventional treatment — The experimental group will receive 5 physiotherapy sessions at home or in a physical therapy office. The respiratory techniques follow a flowchart which begins with saline instillation into the nose and nasopharyngeal cleaning techniques. Then to clear the lung slow inspiratory and slow and forced expiratory techniques will be used. The application of vibration is also included on the flowchart. During the sessions, educational information will also be provided.
  Other Names: Experimental
  Arms: Physiotheraphy + Conventional treatment
Other: Conventional treatment — Medication and observation by a physician/paediatrician. Only evaluations will be made at baseline and on the 3th, 5th and 21st days and an interview 30 days after.
  Other Names: Control
  Arms: Conventional treatment

SUMMARY:
This study aims to evaluate the recovery of children with bronchiolitis with and without physical therapy treatments.

The experimental group will receive educational information and 5 sessions of physiotherapy with the same protocol, at home or in physical therapy office. The control group will only be evaluated.

For both the experimental and control groups the lung sounds are recorded and the Wang's respiratory severity scale calculated initially and on the 3th, 5th and 21st days and computorized. After 3 months of the initial contact, there will be an interview by the phone about relapses or other clinical signs of bronchiolitis until then.

It is expected that the children receiving physiotherapy have a better recovery than the control group.

DETAILED DESCRIPTION:
Due to different opinions in the literature about the relevance of respiratory physiotherapy in the treatment of bronchiolitis, there is an urgent need to conduct studies with robust methodologies to explore the impact of physical therapy in children with bronchiolitis, especially on non-hospitalized, and to consider the different levels of severity of bronchiolitis.

This study aims to evaluate the recovery of children with bronchiolitis with and without physical therapy treatments primarily through the computerized respiratory sounds. As secondary goals secondary measures will be registered to evaluate and compare treatments, such as the duration and frequency of bronchiolitis until 3 months after the diagnosis.

The plan is to recruit approximately 52 children (until the age of 2) with 1st or 2nd bronchiolitis diagnostic by a pediatrician.

Then, the researcher will contact the legal representative of the participants to provide more detailed information and obtain the consent forms. Patients will then be randomly assigned to the conventional treatment group or the conventional treatment plus respiratory physiotherapy group.

The experimental group will receive 5 physiotherapy sessions at home or in a physical therapy office. The respiratory techniques follow a flowchart wich begins with saline instillation in the nose and nasopharyngeal cleaning techniques. Then to clear the lung slow inspiratory and slow and forced expiratory techniques will be used. The application of vibration is also included on the flowchart. During the sessions, educational information will also be provided.

The baseline evaluation will include sociodemographic, anthropometric and clinical data, the calculation of Wang's score and well as computerized lung auscultation. The lung sounds are recorded on 7 anatomic regions: trachea (sternum node) left and right anterior regions (middle clavicular line over the 2nd intercostal space), left and right lateral regions (axillary line over the 4th / 5th intercostal space), left and right back regions (5 cm from the para-vertebral line and 7 cm under the inferior angle of scapular) for approximately 20 seconds.

With the exception of the sample characterization data to be retrieved only in the first evaluation, all other measures will take place in the remaining three evaluations (3th, 5th and 21st days).

The experimental group will still have a final evaluation (auscultation, vital signs and Wang scale) at the end of each treatment session.

A follow-up evaluation will take place after 3 months with a phone interview regarding questioning the recurrence of bronchiolitis, as well as the current presence of symptoms such as cough, sore throat, nasal obstruction, respiratory noise, difficulty sleeping or feeding At the end of this study are expected better results on the experimental group, based on a robust methodology on the impact of respiratory therapy in children from 0 to 2 years, on the treatment bronchiolitis in order to justify the intervention of physiotherapy in this area and to generate recommendations for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* medical diagnostic for 1st or 2nd episode of bronchiolitis and were healthy three days before the current diagnosis of bronchiolitis

Exclusion Criteria:

* comorbidities that can aggravate the severity of bronchiolitis (such as congenital heart disease, Down syndrome, immunosuppression due to medication or diagnosed disease, cystic fibrosis, among others)
* musculoskeletal disorders (eg, scoliosis) and neurological (eg, cerebral palsy) that can interfere with data collection and analysis..

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Computerized lung sounds | From the 1st to the 21st day.
  Adventitious lung sounds are sounds superimposed on the normal respiratory sound. There are continuous (wheezes) and discontinuous (crackles) adventitious sounds. They will indicate the severity and recovery of lung disease

SECONDARY OUTCOMES:
Wang severity scale | From the 1st to the 21st day.
  Classification of severity of respiratory condition by Wang scale through the respiratory rate, presence of wheezing, retractions and overview.

CONTACTS AND LOCATIONS:
Overall Officials: Alda M Marques, PhD, Study Chair — Aveiro University; Veronica L Abreu, MsH, Principal Investigator — Universidade do Porto; José A Duarte, PhD, Study Chair — Universidade do Porto
Locations (1):
- Faculdade de Desporto da Universidade do Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marques A, Oliveira A, Jacome C. Computerized adventitious respiratory sounds as outcome measures for respiratory therapy: a systematic review. Respir Care. 2014 May;59(5):765-76. doi: 10.4187/respcare.02765. Epub 2013 Sep 17. PMID 24046460
- [Derived] Roque-Figuls M, Gine-Garriga M, Granados Rugeles C, Perrotta C, Vilaro J. Chest physiotherapy for acute bronchiolitis in paediatric patients between 0 and 24 months old. Cochrane Database Syst Rev. 2023 Apr 3;4(4):CD004873. doi: 10.1002/14651858.CD004873.pub6. PMID 37010196